CLINICAL TRIAL: NCT04415541
Title: Psychodynamic Psychotherapy for Psychosis: An Empirical Pilot Study of Efficacy, Therapeutic Action, and Machine Learning Analysis of Within-Session Speech and Behavior
Brief Title: Psychodynamic Psychotherapy for Psychosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID
Sponsor: Yale University (Other)
Collaborators: University of Southern California (Other); American Psychoanalytic Association (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000028087
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Psychotic Disorders
MeSH Terms: conditions — Psychotic Disorders | interventions — Psychotherapy, Psychodynamic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychodynamic Psychotheray (Experimental): Following Coordinated Specialty Care, we will offer weekly psychodynamic psychotherapy and medication management sessions which will be conducted solely by the PI, Keith Gallagher, in the initial pilot period. Consent will be obtained to record audio and video of the sessions
  Interventions: Behavioral: Psychodynamic Psychotherapy
- Treatment as Usual (Active Comparator): Following Coordinated Specialty Care, patients will be referred to general mental health providers in the community, which would typically include less intensive and frequent psychotherapy by a social worker or psychologist as well as medication management by a psychiatrist who may not be a specialist in psychotic disorders.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Psychodynamic Psychotherapy — Intensive psychotherapy that is psychodynamically oriented.
  Arms: Psychodynamic Psychotheray
Behavioral: Usual Care — Conventional treatment offered in the community.
  Arms: Treatment as Usual

SUMMARY:
The broad goals of our pilot study are to (1) determine whether psychodynamic psychotherapy for psychosis (PPfP), relative to treatment as usual (TaU), can maintain or augment clinical and functional benefits for patients who have achieved initial recovery in our coordinated specialty care (CSC) early psychosis treatment program; (2) to conduct novel empirical study of how various psychodynamic factors may inform candidate selection, mediate therapeutic effects, and influence relational aspects of the therapy; and (3) to conduct a detailed study of how features of therapist and patient speech and behavior influence therapeutic outcomes, therapeutic alliance alliance, and relational process. This registration focuses on the first goal.

ELIGIBILITY:
Inclusion Criteria:

* completed the 2-3 year Coordinated Specialty Care (CSC) program
* judged by present provider to be in an intermediate or advanced phase of recovery
* had first episode of psychosis within the 3 years prior to enrollment

Exclusion Criteria:

* established diagnosis of primary affective disorder, psychosis secondary to substance use or a medical illness
* inability to communicate in English
* eligibility for Department of Developmental Services
* legally mandated to enter treatment.

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Overall Symptom Severity | From enrollment up to 5 years from enrollment.
  The Positive and Negative Symptom Scale (PANSS) will be used. This is a 30 item scale. Each item is measured on a 7-point scale from 1 (absent) to 7 (extreme). Items are summed to obtain an overall score.
Overall Functioning - Social | From enrollment up to 5 years from enrollment.
  The Global Functioning: Social scale will be used, with symptoms rated 1 (most impaired) to 10 (superior functioning).
Overall Functioning - Role | From enrollment up to 5 years from enrollment.
  The Global Functioning: Role scale will be used, with symptoms rated 1 (most impaired) to 10 (superior functioning).

SECONDARY OUTCOMES:
Symptom Severity (Positive Symptoms) | From enrollment up to 5 years from enrollment.
  The positive symptoms subscale of the Positive and Negative Symptom Scale (PANSS) will be used. Each item is measured on a 7-point scale from 1 (absent) to 7 (extreme). Subscale items are summed to obtain a positive symptom score.
Symptom Severity (Negative Symptoms) | From enrollment up to 5 years from enrollment.
  The negative symptoms subscale of the Positive and Negative Symptom Scale (PANSS) will be used. Each item is measured on a 7-point scale from 1 (absent) to 7 (extreme). Subscale items are summed to obtain an overall score.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Gallagher, MD, Principal Investigator — Yale University